CLINICAL TRIAL: NCT02545517
Title: A Phase 3, Open-label, Multicenter Study to Evaluate Long-term Immunogenicity and Boostability of Immune Responses in Adults Who Received Different Primary Vaccination Regimens of Pre-exposure Prophylaxis With Purified Chick-Embryo Cell Rabies Vaccine Administered Concomitantly or Separately From a Japanese Encephalitis Vaccine.
Brief Title: A Phase 3 Clinical Trial to Evaluate Long-term Immunogenicity and Boostability of Purified Chick-Embryo Cell Rabies Vaccine in Adults Following Primary Series of Pre/Exposure Prophylaxis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 205214; 2015-000382-31 (EudraCT Number); V49_23E1 (Other: Novartis)
Record Dates: First submitted 2015-08-31; First posted 2015-09-10 (Estimated); Results first posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Virus Diseases; Rabies
Keywords: Rabies disease; Pre-exposure (PrEP) or post exposure prophylaxis (PEP); Long-term Immunogenicity
MeSH Terms: conditions — Virus Diseases; Rabies | interventions — Blood Specimen Collection

ARMS (3):
- Conv-R/JE Group (Experimental): Participants who completed the Rabies PrEP regimen on days 1, 8 and 29, and Japanese Encephalitis (JE) primary series regimen on days 1 and 29 in the parent study (V49_23) and who received at least one booster dose of purified chick embryo cell culture (PCEC) rabies vaccine in this extension study, if Rabies Virus Neutralizing Antibody (RNVA) concentrations were less than (<)0.5 IU/mL at scheduled visits.
  Interventions: Biological: Rabipur; Procedure: Blood sampling; Biological: Purified Chick-Embryo Cell Rabies Vaccine
- Acc-R/JE Group (Experimental): Participants who completed the Rabies PrEP regimen on days 1, 4 and 8 and JE primary series regimen on days 1 and 8 in the parent study (V49_23) and who received at least one booster dose of PCEC rabies vaccine in this extension study, if RNVA concentrations were <0.5 IU/mL at scheduled visits.
  Interventions: Biological: Rabipur; Procedure: Blood sampling
- Conv-R Group (Experimental): Participants who completed the Rabies PrEP regimen on days 1, 8 and 29 in the parent study (V49_23) and who received at least one booster dose of PCEC rabies vaccine in this extension study, if RNVA concentrations were <0.5 IU/mL at scheduled visits.
  Interventions: Biological: Rabipur; Procedure: Blood sampling

INTERVENTIONS:
Biological: Rabipur — Participants in all the groups received Rabipur vaccine booster dose, administered intramuscularly in the deltoid region of the non-dominant arm.
Procedure: Blood sampling — Blood samples were drawn from all participants at Day 1 and then at subsequent year intervals from extension study Day 1 onwards.
Biological: Purified Chick-Embryo Cell Rabies Vaccine — 1 booster dose of 1.0 mL of Purified Chick-Embryo Cell Rabies Vaccine intramuscular (IM).
  Arms: Conv-R/JE Group

SUMMARY:
The aim of this study is to evaluate the long-term (up to approx.10 years) persistence and to assess the boostability of immune responses in participants who received a primary series of accelerated or conventional rabies PrEP IM regimen.

This product has been transferred to BN. GSK Clinical Study Register is no longer maintained for this study. The most up to date information is available on www.clinicaltrials.gov.

ELIGIBILITY:
Inclusion Criteria:

* All individuals who were randomized to a Rabies primary series vaccination for pre-exposure prophylaxis (PrEP), received the full PrEP regimen and completed the parent trial following study protocol.

Exclusion Criteria:

* Completed the parent study without receiving the full 3 rabies vaccine doses following the assigned pre-exposure prophylaxis regimen.
* History of exposure to suspected or confirmed rabid animal.
* Receipt of rabies immunoglobulins, rabies post exposure prophylaxis following completion of the parent study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- GSK Investigational Site, Vienna, Austria
- Germany (4):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Rostock, Mecklenburg-Vorpommern
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- GSK Investigational Site, Zurich, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Up to 459 participants, who successfully completed rabies pre-exposure prophylaxis (PrEP) regimens in parent study (V49_23) (NCT01662440, EudraCT ID- 2011-005173-23) and did not have protocol deviations which could impact the immunogenicity response (e.g., wrong vaccination) were enrolled in this extension study.
Pre-assignment Details: As prespecified in protocol, Visit 1 in the extension study corresponds to Year 3, i.e. approximately 3 years after completion of rabies primary series in the parent study. Subsequent visits (2,3,4,5,6,7 and 8) occurred at yearly intervals applied after completion of parent study (Year 4, 5, 6, 7, 8, 9 and 10).
Period: Overall Study
Arm/Group | Conv-R/JE Group | Acc-R/JE Group | Conv-R Group
Started | 126 | 157 | 176
Completed | 98 | 123 | 135
Not Completed | 28 | 34 | 41
Not completed — Death | 2 | 2 | 1
Not completed — Lost to Follow-up | 14 | 13 | 17
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Withdrawal by Subject | 5 | 8 | 9
Not completed — Administrative reason | 5 | 6 | 10
Not completed — Other | 2 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conv-R/JE Group | Acc-R/JE Group | Conv-R Group | Total
Number analyzed (Participants) | 126 | 157 | 176 | 459
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 37.9 (13.2) | 38.7 (13.0) | 36.6 (12.8) | 37.7 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 94 | 101 | 256
  Male | 65 | 63 | 75 | 203
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ASIAN | 1 | 0 | 1 | 2
  BLACK OR AFRICAN AMERICAN | 0 | 2 | 0 | 2
  OTHER UNSPECIFIED | 0 | 1 | 2 | 3
  WHITE | 125 | 154 | 173 | 452

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs) After a Booster Dose of Purified Chick Embryo Cell Culture (PCEC) Rabies Vaccine
Description: A SAE is defined as any untoward medical occurrence that at any dose results in one or more of the following: death, is life-threatening, required/prolonged hospitalization, persistent or significant disability/incapacity, congenital anomaly/or birth defect, an important and significant medical event that may not be immediately life threatening or resulting in death or hospitalization but, based upon appropriate medical judgment, may jeopardize the participants or may require intervention to prevent one of the other outcomes listed.
  Safety is assessed as the number of participants reporting SAEs after a booster dose of PCEC rabies vaccine administered in this extension study, if RNVA concentrations were <0.5 IU/mL, following a primary series of accelerated or conventional rabies pre-exposure (PrEP) intramuscular (IM) regimen in the parent study.
Time Frame: From booster vaccination [6 to 9 months after Year 3 (3 years after primary series of vaccination)] up until completion of the safety follow-up period (10 years after primary series of vaccination)
Population: The analysis was performed on the Safety Set which included all enrolled participants who received a booster dose and reported safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | Conv-R/JE Group | Acc-R/JE Group | Conv-R Group
Number analyzed (Participants) | 44 | 47 | 53
Participants | 2 | 0 | 3

2. Primary Outcome: Number of Participants Who Had Their Rabies Virus Neutralizing Antibody (RNVA) Concentrations Drop Below 0.5 International Units (IU) Per Milliliter (mL) Between Day 366 and Year 3
Time Frame: Day 366 to Year 3 (after primary series of vaccination)
Population: The analysis was performed on the Full Analysis Set-2 (FAS-2): long term immunogenicity analysis which included all eligible participants from the V49_23 study enrolled in this extension study and provided immunogenicity data for the specific analysis at the specific timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Conv-R/JE Group | Acc-R/JE Group | Conv-R Group
Number analyzed (Participants) | 96 | 98 | 133
Participants | 1 | 1 | 2

3. Primary Outcome: Number of Participants Who Had Their RNVA Concentrations Drop Below 0.5 IU/mL Between Year 3 and Year 4
Time Frame: Year 3 to Year 4 (after primary series of vaccination)
Population: The analysis was performed on the FAS-2: long term immunogenicity analysis which included all eligible participants from the V49_23 study enrolled in this extension study and provided immunogenicity data for the specific analysis at the specific timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Conv-R/JE Group | Acc-R/JE Group | Conv-R Group
Number analyzed (Participants) | 93 | 92 | 133
Participants | 5 | 5 | 7

4. Primary Outcome: Number of Participants Who Had Their RNVA Concentrations Drop Below 0.5 IU/mL Between Year 4 and Year 5
Time Frame: Year 4 to Year 5 (after primary series of vaccination)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Conv-R/JE Group | Acc-R/JE Group | Conv-R Group
Number analyzed (Participants) | 85 | 84 | 117
Participants | 7 | 0 | 4

5. Primary Outcome: Number of Participants Who Had Their RNVA Concentrations Drop Below 0.5 IU/mL Between Year 5 and Year 6
Time Frame: Year 5 to Year 6 (after primary series of vaccination)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Conv-R/JE Group | Acc-R/JE Group | Conv-R Group
Number analyzed (Participants) | 72 | 83 | 112
Participants | 3 | 2 | 10

6. Primary Outcome: Number of Participants Who Had Their RNVA Concentrations Drop Below 0.5 IU/mL Between Year 6 and Year 7
Time Frame: Year 6 to Year 7 (after primary series of vaccination)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Conv-R/JE Group | Acc-R/JE Group | Conv-R Group
Number analyzed (Participants) | 67 | 78 | 101
Participants | 0 | 2 | 0

7. Primary Outcome: Number of Participants Who Had Their RNVA Concentrations Drop Below 0.5 IU/mL Between Year 7 and Year 8
Time Frame: Year 7 to Year 8 (after primary series of vaccination)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Conv-R/JE Group | Acc-R/JE Group | Conv-R Group
Number analyzed (Participants) | 67 | 74 | 97
Participants | 0 | 0 | 0

8. Primary Outcome: Number of Participants Who Had Their RNVA Concentrations Drop Below 0.5 IU/mL Between Year 8 and Year 9
Time Frame: Year 8 to Year 9 (after primary series of vaccination)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Conv-R/JE Group | Acc-R/JE Group | Conv-R Group
Number analyzed (Participants) | 66 | 72 | 93
Participants | 1 | 0 | 2

9. Primary Outcome: Number of Participants Who Had Their RNVA Concentrations Drop Below 0.5 IU/mL Between Year 9 and Year 10
Time Frame: Year 9 to Year 10 (after primary series of vaccination)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Conv-R/JE Group | Acc-R/JE Group | Conv-R Group
Number analyzed (Participants) | 61 | 69 | 85
Participants | 2 | 0 | 0

10. Primary Outcome: RVNA Antibody Concentrations 7 Days After the Booster Dose
Description: RVNA antibody concentrations were measured in terms of Geometric Mean Concentrations (GMCs) and expressed in IU/mL. The booster dose was administered in this Extension study (conducted from Year 3 to Year 9 after the primary schedule study) only when participants had RVNA concentrations <0.5 IU/mL at the yearly immunogenicity check (i.e., at "Scheduled Clinic Visit"). Booster dose administration occurred at an approximate timepoint between 6 and 9 months from the previous "Scheduled Clinic Visit" during the Years 3 to 9.
Time Frame: At Day 7 after booster dose
Population: Analysis was performed on the Full Analysis Set-1 (FAS-1): booster immunogenicity analysis, which included all eligible participants from the V49_23 study enrolled in this extension study, whom received booster dose (booster dose was administered only when participants reached RVNA concentrations <0.5 IU/mL) and provided immunogenicity data for the specific analysis at the specific timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Conv-R/JE Group | Acc-R/JE Group | Conv-R Group
Number analyzed (Participants) | 43 | 46 | 52
IU/mL | 4.2 [2.8 to 6.4] | 4.2 [2.8 to 6.2] | 4.4 [3.0 to 6.4]

11. Primary Outcome: RVNA Geometric Mean Ratios (GMRs) 7 Days After the Booster Dose Versus Antibody Concentrations Before the Booster Dose
Description: GMR was calculated as ratio of post booster dose RVNA GMCs (7-day post booster dose) to the baseline RVNA GMCs (7 days before booster dose). The booster dose was administered in this Extension study (conducted from Year 3 to Year 9 after the primary schedule study) only when participants had RVNA concentrations <0.5 IU/mL at the yearly immunogenicity check (i.e., at "Scheduled Clinic Visit"). Booster dose administration occurred at an approximate timepoint between 6 and 9 months from the previous "Scheduled Clinic Visit" during the Years 3 to 9.
Time Frame: Day 7 after booster dose compared to baseline (7 days before booster dose)
Population: Analysis was performed on the FAS-1: booster immunogenicity analysis, which included all eligible participants from the V49_23 study enrolled in this extension study, whom received booster dose (booster dose was administered only when participants reached RVNA concentrations <0.5 IU/mL) and provided immunogenicity data for the specific analysis at the specific timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Conv-R/JE Group | Acc-R/JE Group | Conv-R Group
Number analyzed (Participants) | 43 | 46 | 52
Ratio | 23.6 [16.1 to 34.4] | 23.4 [16.2 to 33.8] | 19.3 [13.7 to 27.3]

12. Primary Outcome: Percentage of Participants With RVNA Concentrations Greater Than or Equal to (>=) 0.5 IU/mL, 7 Days After Booster Dose
Description: The booster dose was administered in this Extension study (conducted from Year 3 to Year 9 after the primary schedule study) only when participants had RVNA concentrations <0.5 IU/mL at the yearly immunogenicity check (i.e., at "Scheduled Clinic Visit"). Booster dose administration occurred at an approximate timepoint between 6 and 9 months from the previous "Scheduled Clinic Visit" during the Years 3 to 9.
Time Frame: At Day 7 after booster dose
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Conv-R/JE Group | Acc-R/JE Group | Conv-R Group
Number analyzed (Participants) | 43 | 46 | 52
Percentage of participants | 95.3 [84.2 to 99.4] | 89.1 [76.4 to 96.4] | 98.1 [89.7 to 100.0]

13. Primary Outcome: Percentage of Participants With RVNA Concentrations >= 0.5 IU/mL at Year 3
Time Frame: At Year 3 after primary series of vaccine administration
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Conv-R/JE Group | Acc-R/JE Group | Conv-R Group
Number analyzed (Participants) | 125 | 151 | 172
Percentage of participants | 81.6 [73.7 to 88.0] | 78.8 [71.4 to 85.0] | 84.9 [78.6 to 89.9]

14. Primary Outcome: Percentage of Participants With RVNA Concentrations >= 0.5 IU/mL at Year 4
Time Frame: At Year 4 after primary series of vaccine administration
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Conv-R/JE Group | Acc-R/JE Group | Conv-R Group
Number analyzed (Participants) | 121 | 144 | 166
Percentage of participants | 74.4 [65.6 to 81.9] | 70.8 [62.7 to 78.1] | 76.5 [69.3 to 82.7]

15. Primary Outcome: Percentage of Participants With RVNA Concentrations >= 0.5 IU/mL at Year 5
Time Frame: At Year 5 after primary series of vaccine administration
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Conv-R/JE Group | Acc-R/JE Group | Conv-R Group
Number analyzed (Participants) | 118 | 139 | 160
Percentage of participants | 66.1 [56.8 to 74.6] | 69.1 [60.7 to 76.6] | 73.1 [65.6 to 79.8]

16. Primary Outcome: Percentage of Participants With RVNA Concentrations >= 0.5 IU/mL at Year 6
Time Frame: At Year 6 after primary series of vaccine administration
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Conv-R/JE Group | Acc-R/JE Group | Conv-R Group
Number analyzed (Participants) | 110 | 139 | 158
Percentage of participants | 60.9 [51.1 to 70.1] | 66.2 [57.7 to 74.0] | 66.5 [58.5 to 73.8]

17. Primary Outcome: Percentage of Participants With RVNA Concentrations >= 0.5 IU/mL at Year 7
Time Frame: At Year 7 after primary series of vaccine administration
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Conv-R/JE Group | Acc-R/JE Group | Conv-R Group
Number analyzed (Participants) | 108 | 135 | 156
Percentage of participants | 60.2 [50.3 to 69.5] | 64.4 [55.8 to 72.5] | 67.3 [59.3 to 74.6]

18. Primary Outcome: Percentage of Participants With RVNA Concentrations >= 0.5 IU/mL at Year 8
Time Frame: At Year 8 after primary series of vaccine administration
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Conv-R/JE Group | Acc-R/JE Group | Conv-R Group
Number analyzed (Participants) | 107 | 131 | 144
Percentage of participants | 59.8 [49.9 to 69.2] | 64.1 [55.3 to 72.3] | 64.6 [56.2 to 72.4]

19. Primary Outcome: Percentage of Participants With RVNA Concentrations >= 0.5 IU/mL at Year 9
Time Frame: At Year 9 after primary series of vaccine administration
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Conv-R/JE Group | Acc-R/JE Group | Conv-R Group
Number analyzed (Participants) | 108 | 132 | 150
Percentage of participants | 59.3 [49.4 to 68.6] | 63.6 [54.8 to 71.8] | 64.0 [55.8 to 71.7]

20. Primary Outcome: Percentage of Participants With RVNA Concentrations >= 0.5 IU/mL at Year 10
Time Frame: At Year 10 after primary series of vaccine administration
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Conv-R/JE Group | Acc-R/JE Group | Conv-R Group
Number analyzed (Participants) | 105 | 130 | 142
Percentage of participants | 56.2 [46.2 to 65.9] | 62.3 [53.4 to 70.7] | 62.7 [54.2 to 70.6]

21. Secondary Outcome: Rabies Virus Neutralizing Antibody Concentrations
Description: Antibody concentrations were measured in terms of GMCs and expressed in IU/mL.
Time Frame: At Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and Year 10 after primary series of vaccine administration
Population: The analysis was performed on the FAS-2: long term immunogenicity analysis which included all eligible participants from the V49_23 study enrolled in this extension study and provided immunogenicity data for the specific analysis at the specific timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Conv-R/JE Group | Acc-R/JE Group | Conv-R Group
Number analyzed (Participants) | 125 | 151 | 172
IU/mL
  Year 3 | 1.21 [0.88 to 1.65] | 1.16 [0.87 to 1.55] | 1.3 [0.99 to 1.7]
  Year 4: number analyzed (Participants) | 121 | 144 | 166
  Year 4 | 0.69 [0.5 to 0.94] | 0.73 [0.55 to 0.97] | 0.82 [0.63 to 1.07]
  Year 5: number analyzed (Participants) | 118 | 139 | 160
  Year 5 | 0.66 [0.48 to 0.9] | 0.7 [0.53 to 0.94] | 0.74 [0.56 to 0.96]
  Year 6: number analyzed (Participants) | 110 | 139 | 158
  Year 6 | 0.5 [0.37 to 0.69] | 0.6 [0.45 to 0.8] | 0.58 [0.44 to 0.76]
  Year 7: number analyzed (Participants) | 108 | 135 | 156
  Year 7 | 0.49 [0.36 to 0.67] | 0.6 [0.45 to 0.79] | 0.61 [0.47 to 0.8]
  Year 8: number analyzed (Participants) | 107 | 131 | 144
  Year 8 | 0.56 [0.41 to 0.77] | 0.76 [0.57 to 1.01] | 0.68 [0.52 to 0.89]
  Year 9: number analyzed (Participants) | 108 | 132 | 150
  Year 9 | 0.53 [0.39 to 0.73] | 0.7 [0.53 to 0.94] | 0.62 [0.47 to 0.81]
  Year 10: number analyzed (Participants) | 105 | 130 | 142
  Year 10 | 0.59 [0.43 to 0.81] | 0.72 [0.54 to 0.96] | 0.68 [0.52 to 0.89]

22. Secondary Outcome: Reverse Cumulative Percentage for Participants With RVNA Concentrations >=0.5 IU/mL
Description: As specified in the statistical analysis plan, a graphical presentation of the Reverse Cumulative Distribution Plots for participants with RVNA concentrations >=0.5 IU/mL was analyzed for this outcome measure. Due to system constrains, only the reverse cumulative percentage values were reported, to depict the Reverse Cumulative Distribution Plots.
Time Frame: At Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and Year 10 after primary series of vaccine administration
Population: as for outcome 21
Measure: Number; unit: Cumulative percentage of participants
Arm/Group | Conv-R/JE Group | Acc-R/JE Group | Conv-R Group
Number analyzed (Participants) | 125 | 151 | 172
Cumulative percentage of participants
  Year 3 | 100 | 100 | 100
  Year 4: number analyzed (Participants) | 121 | 144 | 166
  Year 4 | 83 | 84 | 83
  Year 5: number analyzed (Participants) | 118 | 139 | 160
  Year 5 | 67 | 70 | 69
  Year 6: number analyzed (Participants) | 110 | 139 | 158
  Year 6 | 54 | 57 | 56
  Year 7: number analyzed (Participants) | 108 | 135 | 156
  Year 7 | 43 | 45 | 44
  Year 8: number analyzed (Participants) | 107 | 131 | 144
  Year 8 | 32 | 33 | 32
  Year 9: number analyzed (Participants) | 108 | 132 | 150
  Year 9 | 21 | 22 | 21
  Year 10: number analyzed (Participants) | 105 | 130 | 142
  Year 10 | 10 | 11 | 10

ADVERSE EVENTS:
Time Frame: All Cause Mortality: from Year 3 (3 years after primary series of vaccination) up until completion of the safety follow-up period (10 years after primary series of vaccination) SAEs: from booster vaccination [6 to 9 months after Year 3 (3 years after primary series of vaccination)] up until completion of the safety follow-up period (10 years after primary series of vaccination)
Description: SAEs were collected only from participants who received booster dose. Five deaths were recorded during this extension study but only one of them was reported as SAE as this was the only one that occurred in a participant who received a booster dose. Solicited and non-serious unsolicited AEs were not collected in this study.
Arm/Group | Conv-R/JE Group | Acc-R/JE Group | Conv-R Group
All-Cause Mortality (participants affected / at risk) | 2/126 | 2/157 | 1/176
Serious Adverse Events (participants affected / at risk) | 2/44 | 0/47 | 3/53
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conv-R/JE Group (N=44) | Acc-R/JE Group (N=47) | Conv-R Group (N=53)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/17/NCT02545517/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT02545517/SAP_001.pdf